CLINICAL TRIAL: NCT05921136
Title: Recycling Potential in Endoscopy
Brief Title: Recycling Potential in Endoscopy - a Multicentre Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Georg Dultz, Goethe University Hospital Frankfurt, Johann Wolfgang Goethe University Hospital
Other Study IDs: Flomi
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Sustainable Development
Keywords: endoscopic procedures; endoscopy; environmental health

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present trial is an observational prospective trial. The aim of the present study is to analyse the recycling potential in endoscopy units in hospitals and outpatient facilities. For this purpose, waste is collected for four weeks each at four locations (two inpatient and two outpatient facilities). Questions such as quantity and quality of garbage will be addressed and compared between the different facilities.

DETAILED DESCRIPTION:
Current considerations by various professional societies are developing theoretical concepts with the goal of greenhouse-neutral endoscopy operation. However, the scientific data situation here is expandable. One study calculated an extrapolation for the US based on the mean value of weight and volume of a total of 278 endoscopies in five days at two hospitals. However, a differentiated consideration of various parameters such as examination type and the location of the endoscopy (outpatient vs. inpatient) was missing here.

In different endoscopic departments waste will be weighed. Those are two hospitals (university and non-university) and two outpatient endoscopy units, each for four weeks. The waste will be divided into residual waste, paper and plastic in order to record the possible recycling potential. In addition, it will be investigated how great the savings potential is by avoiding disposable products (gowns, endoscopes).

The present study addresses the following end points:

* Parts of waste per examination in g (residual waste, plastic, paper).
* Savings potential through reusable items (e.g. gowns)
* Comparison of disposable vs. reusable endoscopes
* Descriptive description of the amount of waste at the different locations
* Statistical comparison of the amount of waste in the different locations
* Statistical comparison of the amount of waste per examination
* Statistical comparison of the amount of waste between out-patient and in-patient

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic examination (gastroscopy, colonoscopy, combined gastro and colonoscopy, ERCP, EUS, bronchoscopy)
* Type of examination (interventional vs diagnostic)
* Known multi-resistant germs (yes vs no)

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No patients will be included but only the garbage after the procedures unrelated to patients.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Amount of waste generated per examination in grams (g) | 16 weeks
  The amount of waste per procedure will be collected by weighing the garbage of after every procedure.

SECONDARY OUTCOMES:
Parts of waste per examination in g (residual waste, plastic, paper). | 16 weeks
Saving potential defined by the amount of reusable items in g per procedure (e.g. gowns) | 16 weeks
  The saving potential is defined as the amount of reusable items in g per procedure. Ruasable items are defined as items that are available as one way and multi-way products. An example are gowns.
Comparison of the amount of waste in g in disposable vs. reusable endoscopes. | 16 weeks
Descriptive description of the amount of waste after 4 weeks in kg and per produre in g at the different locations. | 16 weeks
Statistical comparison of the amount of waste in the different locations | 16 weeks
Statistical comparison of the amount of waste per examination | 16 weeks
Statistical comparison of the amount of waste between out-patient and in-patient departments | 16 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - MDZ Magendarmzentrum, Gastroenterologisch, internistische Gemeinschaftspraxis, Darmstadt, Hesse
  - Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Hesse
  - IPG Hanau, Praxis für Gastroenterologie, Hanau, Hesse
  - Klinikum Hanau, Klinik für Gastroenterologie, Diabetologie und Infektiologie, Hanau, Hesse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez de Santiago E, Dinis-Ribeiro M, Pohl H, Agrawal D, Arvanitakis M, Baddeley R, Bak E, Bhandari P, Bretthauer M, Burga P, Donnelly L, Eickhoff A, Hayee B, Kaminski MF, Karlovic K, Lorenzo-Zuniga V, Pellise M, Pioche M, Siau K, Siersema PD, Stableforth W, Tham TC, Triantafyllou K, Tringali A, Veitch A, Voiosu AM, Webster GJ, Vienne A, Beilenhoff U, Bisschops R, Hassan C, Gralnek IM, Messmann H. Reducing the environmental footprint of gastrointestinal endoscopy: European Society of Gastrointestinal Endoscopy (ESGE) and European Society of Gastroenterology and Endoscopy Nurses and Associates (ESGENA) Position Statement. Endoscopy. 2022 Aug;54(8):797-826. doi: 10.1055/a-1859-3726. Epub 2022 Jul 8. PMID 35803275
- [Background] Namburar S, von Renteln D, Damianos J, Bradish L, Barrett J, Aguilera-Fish A, Cushman-Roisin B, Pohl H. Estimating the environmental impact of disposable endoscopic equipment and endoscopes. Gut. 2022 Jul;71(7):1326-1331. doi: 10.1136/gutjnl-2021-324729. Epub 2021 Dec 1. PMID 34853058
- [Derived] Welsch L, Friedrich-Rust M, Tal A, Haider N, Kim S, Schneider M, Schmitt L, Wittersheim L, Schmitt S, Heide A, Heilani M, Zeuzem S, Eickhoff A, Michael FA. Cutting waste in endoscopy: a multicentre observational study in the German healthcare system. Gut. 2025 Nov 10;74(12):1989-1994. doi: 10.1136/gutjnl-2024-333401. PMID 40473397